CLINICAL TRIAL: NCT07046936
Title: The Role of Mitochondrial Bioenergetics in Resilience in Older Adults With Gynecologic Cancer Receiving Cancer Reductive Treatment
Brief Title: Role of Mitochondrial Bioenergetics in Resilience for Gynecologic Cancer
Acronym: MITO-RES
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00128756; ONC-GYN-2402 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-06-05; First posted 2025-07-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gynecologycal Cancer
Keywords: Mitochondrial Bioenergetics; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMCs and muscle biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced gynecological cancers: Participants 50 years and older with suspected or newly diagnosed advanced gynecological cancer (ovarian/primary peritoneal/fallopian tube or endometrial carcinoma of any histological subtype) who are planned to undergo SOC treatment.
  Interventions: Diagnostic Test: muscle sample; Other: blood draw

INTERVENTIONS:
Diagnostic Test: muscle sample — For participants undergoing standard of care interval cytoreductive surgery via laparotomy, a skeletal muscle biopsy from the rectus abdominis muscle (1 cm x 1 cm x 1 cm, ~300 mg) will be collected.
  For participants who undergo standard of care interval cytoreductive surgery with a laparoscopic approach, a skeletal muscle biopsy will be taken from either the rectus abdominis (1 cm x 1 cm x 1 cm, ~300 mg) or the psoas (1 cm x 0.5 cm x 0.5 cm, ~200 mg) muscle.
Other: blood draw — A total of approximately 60mL or 4 tablespoons of blood will be collected throughout the study

SUMMARY:
The purpose of this research study is to see if patients with endometrial and ovarian cancer are willing to complete physical and cognitive assessments before treatment and again after treatment has ended.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, pilot study that is designed to determine the feasibility of assessing resilience in participants 50 years or older with newly diagnosed advanced endometrial or ovarian cancer who are undergoing tumor reduction surgery and chemotherapy. The study will include pre and post treatment measures of physical and cognitive resiliency such as the Short Physical Performance Battery (SPPB),12 Edmonton Symptom Assessment System Revised (ESAS-r),13 and handgrip strength, International Cognitive Cancer Task Force (ICCTF) Battery14 and the Naming Test from the Neuropsychological Assessment Battery (NAB).

In addition, blood and muscle tissues will be collected at baseline and at the time of surgery, respectively for correlative studies to measure mitochondrial respiration.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an IRB-approved informed consent
* Age ≥50 years at the time of enrollment
* Newly diagnosed or suspected FIGO Stage II-IV ovarian/primary peritoneal/fallopian tube carcinoma of any histological subtype OR FIGO Stage II-IV endometrial carcinoma of any histological subtype
* Planned, standard of care treatment consisting of neoadjuvant chemotherapy, tumor reduction surgery, and adjuvant chemotherapy
* Ability to read and understand the English language

Exclusion Criteria:

* Previously treated for ovarian or endometrial cancer
* History of brain metastases, whole brain irradiation, poorly controlled psychiatric disorders defined by hospitalization within the last 3 months for psychiatric diagnoses, traumatic brain injury, cerebrovascular event, or dementia
* Currently taking anti-amyloid agents, cholinesterase inhibitors, or glutamate regulator
* Documented physical or psychological comorbidity that would limit participant's ability to understand or comply with study procedures for the entire length of the study

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a suspected or confirmed diagnosis of ovarian, primary peritoneal, fallopian tube, or endometrial cancer with planned standard of care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Screening rate | Screening
  Proportion of approached patients who signed consent out of the total number of patients who were approached
Enrollment rate | Screening and pretreatment
  Proportion of consented participants who initiated at least one pretreatment assessment or had pretreatment blood drawn out of the total number of consented participants
Completion rate | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy.
  Proportion of enrolled participants who completed at least one posttreatment assessment (cognitive or physical) out of the total number of enrolled participants
Study Feasibility | Screening and up to 30 days following the completion of adjuvant chemotherapy
  ≥80% enrollment rate, ≥80% completion rate (30 of 37)

SECONDARY OUTCOMES:
Edmonton Symptom Assessment System - Revised (ESAS-r) | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  The ESAS-r is a tool is widely used and validated to assess nine symptoms, including pain, nausea, depression, anxiety, tiredness, lack of appetite, well-being, shortness of breath, and overall well-being at the time of questionnaire completion.
Short Physical Performance Battery (SPPB) | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  The SPPB is a measure of lower-extremity physical function consisting of three components: walking speed, repeated chair stands, and standing balance in three increasingly difficult positions.
Walking speed | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Walking speed is assessed by asking the participants to walk at their usual pace over a 4-meter course. Walking speed is scored from zero to four, with four indicating the highest level of performance and zero indicating an inability to complete the task.
Repeated chair stands | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  The time to complete the task will be recorded. Repeated chair stands is scored from zero to four, with four indicating the highest level of performance and zero indicating an inability to complete the task.
Standing balance | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  For the test of standing balance, participants are asked to maintain balance in three positions, characterized by a progressive narrowing of the base of support: feet together (side-by-side), the heel of one foot beside the big toe of the other foot (semi-tandem), and the heel of one foot in front of and touching the toes of the other foot (tandem). For each of the three positions, participants are timed to a maximum of 10 seconds. Standing balance is scored from zero to four, with four indicating the highest level of performance and zero indicating an inability to complete the task.
Handgrip strength | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Handgrip strength is a fundamental measure of upper body muscle strength and overall physical fitness.
Hopkins Verbal Learning Test-Revised (HVLT-R) retention score | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Raw scores from the three learning trials are combined into a total recall score. The number of recalled words during the delayed recall portion of the test is the delayed recall score. The retention score (%) is the result of the delayed recall score divided by the highest raw score from learning trial #2 or learning trial #3.
Trail-Making Test (TMT) A | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  TMT-A measures psychomotor speed, visuospatial search, and target-directed motor tracking.
Trail-Making Test (TMT) B | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  TMT-B measures executive functions such as cognitive flexibility and set-shifting.
Controlled Oral Word Association Test (COWAT) from the Multilingual Aphasia Examination (MAE) | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  The COWAT measures the speed of lexical access, which is the ability to retrieve the meaning and pronunciation of a word from one's mental dictionary.
Neuropsychological Assessment Battery (NAB) Naming Test | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Participant is shown 31 color photographs of objects. The participant is allowed 10 seconds to recall the name of each object.
Complex I- and II-induced maximum oxygen consumption rate in PBMC | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Maximum oxygen consumption rates from mitochondrial complexes I and II are measured by adding specific substrates that activate each complex in PBMCs
Complex I- and II-induced maximum oxygen consumption rate in muscle | Cytoreductive Surgery
  Maximum oxygen consumption rates from mitochondrial complexes I and II are measured by adding specific substrates that activate each complex in muscle tissue

OTHER OUTCOMES:
Expression of proteins involved in mitochondrial bioenergetic activities in PBMCs | Pretreatment and up to 30 days following the completion of adjuvant chemotherapy
  Protein expression related to electron transport chain activity-including components of the Krebs cycle, fatty acid oxidation, and antioxidant pathways-was measured using proteomics in PBMCs
Expression of proteins involved in electron transport chain activities in muscle tissue | Cytoreductive Surgery
  Protein expression related to electron transport chain activity-including components of the Krebs cycle, fatty acid oxidation, and antioxidant pathways-was measured using proteomics in muscle tissue

CONTACTS AND LOCATIONS:
Overall Officials: Bumsoo Ahn, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No